CLINICAL TRIAL: NCT04128306
Title: Localizing in the Brain the Areas of Time to Contact Perception During an Awake Surgery
Brief Title: Brain Areas of Time-To-Contact Perception: an Awake Surgery Study
Acronym: BRAIN-TIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/18/0240
Record Dates: First submitted 2019-10-09; First posted 2019-10-16 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Brain Tumors
Keywords: Time to contact estimation; awake brain surgery; brain tumor; cerebral mapping
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient group (Experimental): A total of 120 patients with brain tumors will be divided into our two groups, divided as follows:
  1. In the group Pre-Per, 20 patients will be included by localization of electrical stimulation (60 patients in total). A patient who would be stimulable in two different areas could be included in two different groups.
  2. In the group Pre-End, the subjects will be distributed by localization of the brain tumor, by lobe. A total of 20 participants will be included per lobe, corresponding to the frontal, temporal or parietal lobes (as a reminder, a tumor in the occipital lobe is an exclusion criterion), for a total of 60 participants
  Interventions: Behavioral: Behavioral task; Procedure: Awake surgery; Other: Neurological assessment
- Control group (Active Comparator): A maximum of 120 healthy matched sex and age subjects with patients will also be included
  Interventions: Behavioral: Behavioral task; Other: Neurological assessment

INTERVENTIONS:
Behavioral: Behavioral task — In the task, participants will see an object approaching toward them. During its movement, the object disappears, and the participants have to press a button to indicate when they estimate the object to contact with them. The motion parameters of the ball will be varied. The pre and post-surgery phases will test the participants in a long duration version of the task, approximately 30 minutes. The per surgery phase will be made of a 5 minutes version of the task, and the participants will receive a direct cortical stimulation for 4 seconds, at an intensity of 1 to 10 milliampere (mA), in the premotor ventral area, or posterior parietal cortex or somesthetic associative areas.
Procedure: Awake surgery — The patient is first anesthetized for opening the scalp and skull, then awake. During this waking phase, the surgeon passes a few quick and simple tests to the patient, visual (for example, line bisection), language (for example, repeating a list of words) etc. While doing this task, the neurosurgeon disrupts the functioning of certain brain regions by direct electrical stimulation of the cortex in order to identify the regions whose dysfunction will have an impact on the current task.
  During the operation, the areas involved in the construction of the peri-personal space will be stimulated by direct electrical stimulation, for a duration of 4 seconds at an intensity of 1 to 10 mA. These areas are:
  * Ventral premotor cortex (with the exception of the primary motor cortex controlling the dominant hand, so as not to interfere with the motor response of the patient)
  * Posterior parietal cortex
  * Associative somesthetic areas
  Arms: Patient group
Other: Neurological assessment — The Mini Mental State Evaluation, which generally assesses the cognitive state of an individual through his 6 subtests testing both working memory, episodic and semantic praxies as well as spatio-temporal orientation capacity.
Other: Neurological assessment — The Wechsler Adult Intelligence Scale was selected for two of its subtests: The Subtest Codes checking the processing of information, visuo-constructive abilities but also attention. The subtest Cubes evaluates the capacities of visuospatial and constructive organizations as well as the referencing of the space in relation to the subject.
Other: Neurological assessment — The State-Trait Anxiety Inventory, consisting of two self-administered questionnaires: Questionnaire A, measuring the state of anxiety of the person on the present moment and B measuring anxiety as a character trait of the person
Other: Neurological assessment — The Verbal Fluences test, in its oral version. Categorial and lexical fluences make it possible to quickly realize a possible lack of the word of the person as well as disturbances of working memory or the capacity of inhibition.
Other: Neurological assessment — The board of the Corsi cubes that evaluates the non-verbal visual-spatial working memory of the participants with a reminder location that tests the visuo-spatial notebook and a reminder to who tests the central administrator of the working memory.
Other: Neurological assessment — The neurocognitive naming test was chosen to verify correct access to both semantic memory and lexicon, as well as to test the early visual process of image processing necessary for our task.
Other: Neurological assessment — Benton lines are commonly used to determine possible deficits in the localization of isolated objects or judgment of line direction.
Other: Neurological assessment — The patient will finally pass a depression assessment test, answering Beck's questionnaire.

SUMMARY:
During a brain surgery targeted to remove a brain tumor, the neurosurgeon wakes up the patient to delimit the tumor area exactly, and identify the surrounding areas, to limit the surgery damages. The present project aims at testing the patient in this awake phase to determine the brain areas implied in time to contact (TTC) perception, a function that allows determining the arrival time of moving objects and used in many tasks of our daily life.

DETAILED DESCRIPTION:
Time to contact (TTC) estimation is a major visual function that allows an observer determining the time a moving object will take to reach him. It is however striking to note that the different brain areas supporting this function are not clearly identified, in particular the contribution of non-visual areas that are engaged in the definition of a peri-personal space for the observer. This lack could be fulfilled during a brain surgery experiment. Indeed, in such a surgery, the patient is awakened, and the surgeon apply direct cortical stimulation to de-activate specific brain areas while testing different cognitive function. The failure to succeed in the task indicates that this area is engaged in the cognitive function. The present study therefore will test different brain areas to investigate their respective contribution in the TTC estimation function.

Three groups of participants will be tested, in pre and per surgery phases. After an initial pre-surgery phase, patients for which the tumor does not interfere with the TTC estimation anility will be enrolled in the Pré-Per group, and tested during the brain surgery. Patients for which the pre-test indicates that the TTC estimation is damaged by the tumor, will be tested in pre-surgery phase only, constituting the Pré-End group. Finally, a control group, paired with the patients, will be tested as well.

For the patients, all the testing phases will be achieved during their medical process. The awake surgery is now a well-established technique, currently and usually done at the University Hospital Toulouse, and the present test in the per surgery phase only lasts a couple of minutes, no more than 5 minutes. As such, there is no additional risk carried out in the project.

ELIGIBILITY:
Inclusion Criteria:

For the patients:

* Brain tumor that does not affect the dominant hand motricity. The patient that have a tumor in an area targeted for a cortical stimulation will be automatically enrolled within the Pre-End group.
* Who will agree with all terms and sign the experimental agreement
* Correct or corrected vision, as allowed by the surgery constraints
* With no known oculomotor abnormalities (list of exclusion in Annexe)
* Affiliated to a social security system

For the control group:

* Who will agree with all terms and sign the experimental agreement
* Correct or corrected vision
* With no known oculomotor abnormalities.
* Affiliated to a social security system

Exclusion Criteria:

For the patients:

* Brain tumor located in the occipital area
* Legally protected patient, or with unknown ability to sign the experimental agreement, as determined by the medical team.
* Medical background of neurological diseases of the central nervous system, as Parkinson, Alzheimer, stroke
* Pregnancy

For the control group:

* Legally protected patient, or with unknown ability to sign the experimental agreement, as determined by the medical team.
* Medical background of neurological diseases of the central nervous system, as Parkinson, Alzheimer, stroke
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral mapping | 61 months
  Look at how the cognitive functions of perception of time before contact are attached to brain structures, their communication with other zones, their alteration due to brain tumors for patients with a brain tumor compared to control subjects. The treatment of the study being an awakened awakening as part of the routine care, there is no risk of serious adverse event.
  Brain mapping will be done through neurological examinations which are questionnaires and a risk-free task. All the tasks and all the questionnaires described in the paragraph "arm and intervention" will make it possible to meet this outcome.

SECONDARY OUTCOMES:
Look the implication of other brain areas | 61 months
  Look to see if brain areas other than those targeted for stimulation in awake surgery are stimulated and therefore play a role in estimating time to contact.The treatment of the study being an awakened awakening as part of the routine care, there is no risk of serious adverse event.
  Other brain areas will be define through neurological examinations which are questionnaires and a risk-free task. All the tasks and the questionnaires described in the paragraph "arm and intervention" will make it possible to meet this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Franck-Emmanuel Roux, MD, Principal Investigator — University Hopsital Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No